CLINICAL TRIAL: NCT01307956
Title: A Phase II Study of Neo-adjuvant Therapy With Oxaliplatin, Leucovorin, 5-Fluorouracil, Panitumumab (Vectibix) and Radiation in Patients With Locally Advanced Adenocarcinoma of the Esophagus or Gastroesophageal Junction
Brief Title: Panitumumab, Combination Chemotherapy, & Radiation Therapy in Esophageal or Gastroesophageal Junction Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug manufacturer - Amgen requested study stop, per DSMB observation in POWER trial
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0221-09-FB; NCI-2010-02056 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH)
Record Dates: First submitted 2011-03-01; First posted 2011-03-03 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Esophageal Adenocarcinoma; Stage IIA Esophageal Cancer; Stage IIB Esophageal Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms | interventions — Fluorouracil; dehydroftorafur; Leucovorin; Oxaliplatin; Panitumumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (panitumumab, chemotherapy, radiation) (Experimental): Patients receive panitumumab IV over 1 hour on day 1. Patients also receive oxaliplatin IV and leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours on day 1 (FOLFOX chemotherapy). Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Within 24 hours of the start of chemotherapy, patients undergo radiation therapy 5 days a week for 5.5 weeks. Patients then undergo surgery within 6-8 weeks after completion of radiation therapy. Patients with residual disease receive 4 additional courses of FOLFOX chemotherapy on days 1, 15, 29, and 42.
  Interventions: Drug: Fluorouracil; Other: Laboratory Biomarker Analysis; Drug: Leucovorin Calcium; Drug: Oxaliplatin; Biological: Panitumumab; Other: Pharmacological Study; Radiation: Radiation Therapy; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: Fluorouracil — Given IV
  Other Names: 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; Citrovorum Factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; MoAb ABX-EGF; Monoclonal Antibody ABX-EGF; Vectibix
Other: Pharmacological Study — Correlative studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; Irradiation; RADIATION; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection

SUMMARY:
This phase II trial is studying how well giving panitumumab, combination chemotherapy, and radiation therapy together before surgery works in treating patients with advanced esophageal or gastroesophageal (GE) junction cancer. Monoclonal antibodies, such as panitumumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy x-rays to kill tumor cells. Giving monoclonal antibody therapy together with chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pathologic complete response rate of a modified FOLFOX-6 regimen (leucovorin calcium, fluorouracil, and oxaliplatin) given with panitumumab at two-week intervals x 4 cycles in combination with external beam radiation therapy for patients with locally advanced adenocarcinoma of the esophagus.

SECONDARY OBJECTIVES:

I. To determine the toxicities and ability to complete the planned treatment. II. To determine the achieved steady-state plasma concentrations of 5-FU (fluorouracil) and correlate these with clinical toxicity.

III. To assess the potential importance of polymorphic variations in genomic deoxyribonucleic acid (DNA) of pertinent genes whose protein products are the targets of the anti-neoplastic drugs used in the clinical protocol on response and toxicity to therapy.

OUTLINE:

Patients receive panitumumab intravenously (IV) over 1 hour on day 1. Patients also receive oxaliplatin IV and leucovorin calcium IV over 2 hours, and fluorouracil IV continuously over 46 hours on day 1 (FOLFOX chemotherapy). Treatment repeats every 2 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Within 24 hours of the start of chemotherapy, patients undergo radiation therapy 5 days a week for 5.5 weeks. Patients then undergo surgery within 6-8 weeks after completion of radiation therapy. Patients with residual disease receive 4 additional courses of FOLFOX chemotherapy on days 1, 15, 29, and 42.

After completion of study treatment, patients are followed up every 3 months for 2 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have resectable adenocarcinoma of the esophagus or GE-junction and are medically fit to undergo surgery; patients must have no evidence of distant metastasis based on imaging studies
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) of at least 2000 per mcL
* Platelet count of at least 100,000 per mcL
* Serum creatinine less than or equal to 2.0 mg/dL
* Serum magnesium greater than or equal to 1.8 mg/dL
* Total bilirubin less than or equal to 2.0 mg per dL
* Measurable disease is not required for this study, since the primary endpoint is complete pathologic response
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* Prior therapy: patients with prior history of mediastinal radiation exposure will be ineligible; patients may not have received prior chemotherapy, or antibody therapy for esophageal or GE-junction adenocarcinoma
* History of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Patients with a prior history of marked intolerance to 5-fluoropyrimidines (5-FU, floxuridine, capecitabine, 5-fluorocytosine [flucytosine]), since such patients may have deficiency of dihydropyrimidine dehydrogenase, which places them at risk for severe and life-threatening toxicity with 5-FU
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, ongoing immunosuppressive therapy (except for replacement steroids), active human immunodeficiency virus (HIV) infection, that might jeopardize the ability of the patient to receive the chemotherapy program outlined in this protocol with reasonable safety
* Clinically significant cardiac disease (including symptomatic congestive heart failure, myocardial infarction, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia) within 1 year of study enrollment
* Pregnant and nursing women, or women planning to become pregnant within 6 months after the end of treatment, are excluded from this study; a negative pregnancy test will be required of women of child-bearing age within 72 hours of study enrollment; subjects (male or female) who are not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment are excluded
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest computed tomography (CT) scan
* Patients with prior malignancy will be excluded except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancers from which the patient has been disease-free for at least 5 years
* Patients receiving an investigational agent within 30 days before enrollment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-02-28 (Actual); Primary Completion 2015-12-23 (Actual); Study Completion 2015-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Grem, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10
  Asian/Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathological Response (pCR) Rate
Description: Based on the proportion who achieve pCR based on the first 4 courses of protocol treatment. Evaluated using the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guidelines. Means (with associated standard errors), medians (with ranges), percentages and 95% confidence intervals will be reported as appropriate.
Time Frame: Up to 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Number of Patients Who Can Undergo Resection
Description: Restaging with repeat imaging studies will be performed. If no contraindication for surgical resection is identified, resection will be performed. Means (with associated standard errors), medians (with ranges), percentages and 95% confidence intervals will be reported as appropriate.
Time Frame: 4 weeks after completion of the radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Number analyzed (Participants) | 11
Participants | 11

3. Other Pre Specified Outcome: Progression-free Survival
Description: Descriptively summarized using the method of Kaplan-Meier. Response and disease progression were assessed using RECIST criteria version 1.1
Time Frame: Patients were followed from time of consent until the date of first documented progession or date of death from any cause, whichever came first, assessed up to 100 months.
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Number analyzed (Participants) | 11
days | 409 [119 to 2840]

4. Other Pre Specified Outcome: Overall Survival
Description: Descriptively summarized using the method of Kaplan-Meier.
Time Frame: From the first date of therapy until the date the patient dies, assessed up to 100 months
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
Number analyzed (Participants) | 11
days | 596 [119 to 2840]

ADVERSE EVENTS:
Time Frame: Patients were followed for adverse events from the time of first treatment until they 30 days after last day of study treatment. (approximately 10 weeks)
Arm/Group | Treatment (Panitumumab, Chemotherapy, Radiation)
All-Cause Mortality (participants affected / at risk) | 7/11
Serious Adverse Events (participants affected / at risk) | 10/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panitumumab, Chemotherapy, Radiation) (N=11)
Anemia (Blood and lymphatic system disorders) | 1 (4)
Weight loss (Investigations) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (2) — pulmonary embolism
diarrhea (Gastrointestinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) — deep vein thrombosis
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (6)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 3 (5) — including pneumonia
nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 2 (3)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sepsis (Infections and infestations) | 2 (2)
hypotension (Vascular disorders) | 3 (4)
bradycardia (Cardiac disorders) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — odynophagia
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — melena
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — pneumatosis
Pericarditis (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Surgical and medical procedures - Other (Surgical and medical procedures) | 2 (2) — Tracheotomy
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
alcohol intolerance (Metabolism and nutrition disorders) | 1 (1)
suicidal ideation (Psychiatric disorders) | 1 (1)
hallucinations (Psychiatric disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Troponin increase (Investigations) | 1 (1)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) — abdominal perforation
Typhlitis (Gastrointestinal disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
lymphocyte count decreased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Investigations - Other (Investigations) | 1 (2) — infiltrates
General disorders - Other (General disorders) | 1 (1) — general edema
pain (General disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) — esophageal stricture due to esophagectomy surgery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Panitumumab, Chemotherapy, Radiation) (N=11)
Anorexia (Metabolism and nutrition disorders) | 8 (10)
Hypokalemia (Metabolism and nutrition disorders) | 9 (19)
lymphocyte count decreased (Investigations) | 7 (36)
White blood cells decreased (Investigations) | 8 (18)
Neutrophil count decreased (Investigations) | 7 (13)
Platelet cell count decreased (Investigations) | 2 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (27)
depression (Psychiatric disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 4 (5)
mucositis - oral (Gastrointestinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2) — pneumonia
Acidosis (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (6)
blood bilirubin increased (Investigations) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) — c. difficile
dysgeusia (Nervous system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 4 (5)
Pain (General disorders) | 2 (3)
Hypotension (Vascular disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) — Neurology- sedation
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) — prolonged intubation
INR increased (Investigations) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — pain - knee pain - shoulder
Skin and subcutatneous tissue disorder - Other (Skin and subcutaneous tissue disorders) | 1 (1) — rash
hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (6)
hyponatremia (Metabolism and nutrition disorders) | 1 (2)
Injury, poisoning and procedural complications - Other (Gastrointestinal disorders) | 1 (1) — Esophageal obstruction, stricture at anastomosis
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2)
Alanine aminotransferase (Investigations) | 1 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (1) — jejunal tube clogged, replaced
weight loss (Investigations) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (2)
thromboembolic event (Vascular disorders) | 1 (1) — pulmonary embolism
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 (2) — Pain - chest tube sites
Alkaline phosphatase increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No